CLINICAL TRIAL: NCT06468748
Title: The Effects of a GLP-1R Agonist (the Drug Wegovy®) on Body Composition and Performance in Military Personnel
Brief Title: The Effects of Semaglutide on Body Composition and Performance in Military Personnel
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brandon Roberts, Principal Investigator, United States Army Research Institute of Environmental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-05H
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semaglutide Treatment (Experimental): Semaglutide will be self-administered by participants with a prefilled pen injector on the same day each week, at any time of day, with or without meals. It will be initiated at a dose of 0.25 mg once weekly for the first 4 weeks, with the dose increased every 4 weeks to reach a maintenance dose of 2.4 mg weekly by week 16. They will remain on the maintenance dosage of 2.4mg until week 24. If participants cannot reach 2.4 mg/week they will stop at the maximal tolerable dose (e.g., 1.7 mg/week).
  After 24-weeks, treatment will be stopped, and participants will remain in the trial for 1 year with follow-up assessments at week 48 and week 76.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — During the first visit, participants will be taught how to self-administer the pen injector by medical staff. Participants will also be provided instructions for self-administering injections and a compliance log to track adherence to the treatment, and additional information about each injection (date, time, injection site)

SUMMARY:
The obesity epidemic presents a growing concern in the United States, affecting more than 42% of adults. This epidemic extends its impact to chronic diseases and escalating healthcare expenses. Its reach has even influenced the military, with more than 20% of Soldiers being classified as obese, based on Body Mass Index ≥30 kg/m2. Current preventative and countermeasures have produced limited success, prompting consideration of pharmacotherapy. Within this context, glucagon-like peptide-1 receptor agonists (GLP-1RAs), such as semaglutide, have emerged as a promising treatment for obesity. Semaglutide can induce significant weight loss, primarily through fat reduction. However, questions persist regarding its effects on lean mass, physical performance, bone structure, and how it influences the underlying metabolic and hormonal milieu. Furthermore, no studies have been completed in military personnel, who must exercise regularly. Therefore, the investigators will conduct a single-center, open-label, observational trial. The trial will consist of a 24-week semaglutide treatment period and a non-treated 52-week follow-up period. We will test the feasibility and potential benefits of semaglutide in military populations, with a focus on understanding how semaglutide influences body composition, physical performance, hormones, and metabolism. This research holds military significance as obesity rates among service members continue to rise, undermining their medical readiness. Ultimately, it is important to understand if GLP-1RAs can provide a viable solution to obesity in military personnel and if there might be an unexpected effect on physical readiness due to the nature of the weight loss. This could cut down on healthcare expenses by reducing the reliance on weight-related initiatives and, consequently, lowering military separations.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty military personnel
* Age ≥ 18 years at the time of signing informed consent.
* Body mass index (BMI) ≥ 30 kg/m2 or ≥ 27 kg/m2 with the presence of at least one weight-related comorbid condition (e.g., hypertension, dyslipidemia, etc.)
* History of at least one self-reported effort to lose body weight.
* Ability to exercise ≥ 3x per week during the study.

Exclusion Criteria:

* Currently in Basic Combat Training, Advanced Individual Training, or One Station Unit Training, or equivalence in other military services.
* Current or history of Type 1 or Type 2 Diabetes, cardiovascular (e.g., heart disease, peripheral artery disease), musculoskeletal (e.g., myopathies), immune (e.g., lupus, asthma), gastrointestinal (e.g., irritable bowel syndrome, pancreatitis), neurological (e.g., dystonia), pulmonary (pulmonary fibrosis, COPD, lung cancer), or renal diseases (e.g., kidney diseases), and eating disorders (e.g., bulimia nervosa, anorexia nervosa).
* History of cholecystectomy
* Personal or family history of medullary thyroid carcinoma or those with multiple endocrine neoplasia type 2.
* Participants who are pregnant or breastfeeding, or those who may be pregnant or were pregnant in the last 12 months.
* Male and female participants who plan or will attempt to become pregnant or help conceive a child within two months of treatment.
* Inability to exercise ≥ 3x per week during the study.
* Currently taking or history of routine use of medications known to affect metabolism or performance (e.g., thiazide diuretics, oral steroids, testosterone replacement therapy, etc.).
* Self-reported change in body weight ≥ 5 kg within 90 days before screening.
* Treatment with any medication for the indication of obesity within 90 days before screening.
* Treatment with other orally administered medications such as sulfonylureas, sitagliptin, phenytoin, levothyroxine, albuterol, prednisone, and other drugs as identified during screening by the medical screening and staff.
* Current or previously suspected alcohol abuse (defined as Harmful Use by the World Health Organization), those who meet criteria for alcohol abuse disorder (as outlined in the DSM-5), or other substance abuse (i.e., the use of illegal drugs or the use of prescription or over-the-counter drugs for purposes other than those for which they are meant to be used, or in excessive amounts.
* History of major depressive disorder.
* Participants with implanted or external electrical devices (e.g., pacemakers).
* On a specialized diet (e.g., keto, intermittent fasting).
* Claustrophobia or difficulty breathing with a face mask.
* Known or suspected hypersensitivity to study product(s) or related products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 24 weeks
  the amount of body weight loss in kilograms caused by semaglutide in 24 weeks.
Body composition | 24 weeks
  the percentage of lean and fat mass loss during semaglutide treatment.
Physical Performance | 24 weeks
  the percent change in VO2peak (mL/kg/min) during semaglutide treatment.

SECONDARY OUTCOMES:
Weight Loss Maintenance | 76 weeks
  if semaglutide results in maintenance of lower body weight in kilograms 52 weeks after cessation of treatment.
Eating habits and mediators of eating behavior | 76 weeks
  the effects of semaglutide treatment on appetite, hunger, and food preferences measured by the military eating behavior scale during and after semaglutide treatment.

OTHER OUTCOMES:
Bone | 76 weeks
  the effects of semaglutide treatment on bone volume/total volume during and after semaglutide treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No